CLINICAL TRIAL: NCT03551821
Title: An Open-Label Pilot Study of the Safety, Tolerability and Efficacy of ATI-50002 Topical Solution Administered Twice-Daily in Adult Subjects With Eyebrow Loss Due to Alopecia Areata, Alopecia Universalis or Alopecia Totalis
Brief Title: Open Label Study of ATI-50002 Topical Solution Administered to Adult Subjects With Eyebrow Loss Due to Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI-50002-AAB-201
Record Dates: First submitted 2018-05-17; First posted 2018-06-11 (Actual); Results first posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-10

CONDITIONS: Alopecia Areata; Alopecia Totalis; Alopecia Universalis
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATI-50002 Topical Solution (Experimental): ATI-50002 Topical Solution
  Interventions: Drug: ATI-50002

INTERVENTIONS:
Drug: ATI-50002 — Topical Solution

SUMMARY:
The main objective of this study is to assess the safety, tolerability and efficacy of ATI-50002 Topical Solution in subjects with unilateral or bilateral loss of eyebrow hair due to alopecia areata (AA), alopecia universalis (AU) or alopecia totalis (AT).

DETAILED DESCRIPTION:
This is an open-label study which will be conducted at 1 to 2 sites.

Subjects will be required to have a clinical diagnosis of AA, AU or AT with unilateral or bilateral loss of eyebrow hair.

Subjects will apply study medication to the entire affected eyebrow(s), twice-daily for 24 weeks.

Safety and tolerability will be evaluated throughout the study.

The duration of the study participation is anticipated to be a maximum of 233 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age.
2. Subject has, based on a subject history and clinical examination, a clinical diagnosis of AA, AU or AT with no eyebrow hair in the affected area(s) and no eyebrow regrowth over the previous 6 months. Affected area is defined as the area(s) of eyebrow hair loss identified at Baseline.
3. Subject has a Clinician Eyebrow Assessment score of 0 for at least one eyebrow.
4. Subject has a Subject Eyebrow Assessment score of 0 for at least one eyebrow.
5. Subject has a duration of the current episode of AA, AU or AT with unilateral or bilateral loss of eyebrow hairs (with at least one distinct patch of >30% loss of eyebrow hair) for at least 6 months and no more than seven years prior to Visit 1.
6. Subjects who are Women of Childbearing Potential (WOCBP) must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline and agree to use a highly effective method of birth control for the duration of the study and for 30 days after last study medication application.
7. Subject is non-pregnant and non-lactating and not planning a pregnancy during the duration of the study and for 30 days after the last study medication application.
8. Subject is in good general health and free of any known disease state or physical condition which, in the opinion of the investigator, would interfere with the study requirements or put the subject at undue risk by study participation.
9. Subject is willing and able to follow all study instructions and to attend all study visits.
10. Subjects taking hormonal replacement therapy must have been on the same dose for at least 6 months prior to Visit 1 and must agree to maintain the same dose for the duration of the study and for 90 days after the last study medication application.
11. Subjects taking thyroid replacement therapy must have been on the same dose for at least 6 months prior to Visit 1 and must agree to maintain the same dose for the duration of the study.
12. Subject agrees to refrain from any eyebrow removal (e.g.¸ plucking, threading, etc.) for the duration of the study.
13. Subject agrees to refrain from any cosmetic surgery (e.g., piercing, tattooing, etc.), on the treatment areas, for the duration of the study.
14. Subject can comprehend and is willing to sign an Informed Consent Form (ICF).
15. Sexually active male subjects must agree to use a barrier method of contraception from the first application of study medication to at least 30 days after the last application of study medication

Exclusion Criteria:

1. Subject has, in the opinion of the investigator, permanent eyebrow loss attributed to causes other than AA, AU or AT such as overgrooming, or scarring hair loss.
2. Subject currently has, or has a history of, skin disease in the eyebrow area (e.g., psoriasis, seborrheic dermatitis, etc.) that, in the opinion of the investigator, would interfere with the study medication application or study assessments.
3. Subject currently has, or has a history of, severe, progressive or uncontrolled autoimmune, metabolic, endocrinologic, renal, hepatic, gastrointestinal, pulmonary, cardiovascular, genitourinary (i.e., renal disease), hematological disease, neurologic or cerebral disorders, infectious disease or coagulation disorders that, in the opinion of the investigator, put the subject at undue risk by study participation.
4. Subject currently has, or has a history of, proven or suspected systemic or cutaneous malignancy and /or lymphoproliferative disease, other than a history of adequately treated, well healed and completely cleared non-melanoma skin cancers (e.g. basal or squamous cell carcinoma) treated successfully at least one year prior to Visit 1.
5. Subject currently has evidence of active or latent bacterial infection, including tuberculosis, or viral infections at the time of enrollment or a history of incompletely treated or untreated tuberculosis. Subjects who have completed therapy for latent tuberculosis may participate.
6. Subject has a history of serious local infection (e.g., cellulitis, abscess) or a systemic infection, including but not limited to, pneumonia or septicemia, within 12 weeks prior to Visit 1. Subjects on an antibiotic for a nonserious, acute local infection must complete the antibiotic course prior to enrollment in the study.
7. Subjects positive for HIV, Hepatitis B or C.
8. Subject currently has or has a known history of herpes zoster or cytomegalovirus (CMV) within 8 weeks prior to Visit 1.
9. Subject has a history of frequent outbreaks of Herpes Simplex Virus defined as 4 or more episodes per year.
10. Subject has any history of eyebrow tattooing, or microblading that in the opinion of the investigator would interfere with the assessment of safety or efficacy.
11. Subject has used any semi-permanent eyebrow coloring (e.g., tinting, dying, etc.) within 6 months prior to Visit 1 that in the opinion of the investigator would interfere with the assessment of safety or efficacy.
12. Clinically significant laboratory abnormalities at Screening that, in the opinion of the Investigator, would make the subject a poor candidate for the study.
13. Subjects with absolute neutrophil count <1,000/mm3, or platelet count <50,000/ml.
14. Subject used any of the following therapies within the specified period prior to Visit 1:

    Systemic therapies:
    * Disease Modifying Anti-Rheumatic Drugs (DMARDS), Biologics or immunosuppressants, such as: anakinra, adalimumab, azathioprine, glucocorticosteroids, cyclosporine, etanercept, infliximab, methotrexate, TNF inhibitors, ustekinumab, secukinumab, ixekizumab, certolizumab pegol: 4 weeks or 5 half-lives whichever is longer
    * Oral retinoids: 12 weeks
    * Plaquenil: 8 weeks
    * JAK inhibitors (oral or topical): 1 year
    * Intralesional steroids on the eyebrow area: 4 weeks

    Topical therapies on the eyebrow area:
    * Phototherapy, Laser Therapy : 12 weeks
    * Anthralin, bimatoprost, glucocorticosteroids, diphencyprone, diphenylcycloprophenone (DPCP), Squaric acid dibutyl ester (SADBE), minoxidil, pimecrolimus, tacrolimus: 4 weeks
    * Topical treatments (prescription and over-the-counter) that contain retinoids, retinol, alpha hydroxy acids (e.g. glycolic, lactic acids) and beta hydroxy acids (e.g. salicylic acid) on and around the eyebrow area: 4 weeks
15. Subject has a history of sensitivity to any of the ingredients in the study medication.
16. Subject has participated in an investigational drug or device trial in which administration of an investigational study drug or device occurred within 30 days or 5 half-lives (whichever is longer) prior to Visit 1. Subjects who have participated in a study of an investigational drug, device or biologic agent for alopecia areata (AA, AU or AT) within 1 year of screening will be eligible to participate only with individual permission from the Medical Monitor.
17. History of or current alcohol or drug abuse within 2 years of assessment for study enrollment.
18. Screening ECG findings of:

    * QTcF >450msec for males or >470msec for females (use of the ECG algorithm is acceptable for this purpose)
    * Heart rate < 45 or > 100 beats/minutes (inclusive)
    * Rhythm disturbance other than sinus arrhythmia or ectopic supraventricular rhythm (ectopic atrial rhythm)
    * Conduction disturbance including PR >240msec, pre-excitation (delta wave and PR <120msec), second degree or higher AV block
    * Acute or chronic signs of ischemia
    * Left Bundle Branch Block
    * Prior myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Aclaris Investigator Site, Boynton Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ATI-50002 Topical Solution
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 50 [50 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinician's Eyebrow Assessment
Description: Determination of the amount of hair in the affected area.
  Clinician's Eyebrow Assessment
  Grade Descriptor 0 No eyebrow hair: No terminal hairs are visible in the affected area(s)
  1. A little eyebrow hair: Occasional terminal hairs are visible in the affected area(s)
  2. Some eyebrow hair: Numerous terminal hairs are visible in the affected area(s)
  3. Most eyebrow hair: Mostly complete eyebrow regrowth with terminal hair in the affected area(s)
  4. Full eyebrow hair: Complete eyebrow regrowth with terminal hair in the affected area(s)
Time Frame: Six months
Measure: Number; unit: score on a scale
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 1
score on a scale | 0

2. Secondary Outcome: Subject's Eyebrow Assessment
Description: Determination of the amount of hair in the affected area.
  Subject's Eyebrow Assessment Grade Descriptor 0 No eyebrow hair: No thick, coarse hairs are visible in the affected area(s)
  1. A little eyebrow hair: A few thick, coarse hairs are visible in the affected area(s)
  2. Some eyebrow hair: Numerous thick, coarse hairs are visible in the affected area(s)
  3. Most eyebrow hair: The majority of the affected area(s) of the eyebrow is covered in thick, coarse hairs
  4. Full eyebrow hair: The affected area(s) of the eyebrow is fully covered in thick, coarse hairs
Time Frame: Six months
Measure: Number; unit: score on a scale
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 1
score on a scale | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | ATI-50002 Topical Solution
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT03551821/Prot_SAP_000.pdf